CLINICAL TRIAL: NCT06350825
Title: Evaluating the Efficacy and Safety of Cytoreductive Prostatectomy Combined With Triple or Dual Systemic Therapy in Patients With Metastatic Hormone-Sensitive Prostate Cancer
Brief Title: Cytoreductive Prostatectomy Combined With Triple or Dual Systemic Therapy in mHSPC Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hua Lixin, Clinical Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SR-543
Record Dates: First submitted 2024-03-20; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Prostate Cancer; Therapy, Directly Observed
Keywords: prostate cancer; cytoreductive prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms; Directly Observed Therapy | interventions — Brachytherapy; Surgical Procedures, Operative; Drug Therapy

STUDY DESIGN:
Intervention Model Description: randomized control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local treatment group (Experimental): Triplet or doublet therapy followed by cytoreductive prostatectomy or brachytherapy
  Interventions: Procedure: Cytoreductive prostatectomy or brachytherapy
- SOC group (Active Comparator): Triplet or doublet therapy (ie. docetaxel/abiraterone, apalutamide，Rezvilutamide，darolutamide，enzalutamide)
  Interventions: Drug: ADT+second-generation antiandrogens ± chemotherapy

INTERVENTIONS:
Procedure: Cytoreductive prostatectomy or brachytherapy — local treatment+SOC for metastatic prostate cancer
  Other Names: surgery or radiation therapy+SOC
  Arms: Local treatment group
Drug: ADT+second-generation antiandrogens ± chemotherapy — SOC(Triplet or doublet therapy) for mHSPC
  Other Names: hormonal therapy or chemotherapy
  Arms: SOC group

SUMMARY:
To evaluate: The radiographic progression-free survival (rPFS) of metastatic hormone-sensitive prostate cancer (mHSPC) patients treated with androgen deprivation therapy (ADT) + second-generation antiandrogens±chemotherapy combined with cytoreductive prostatectomy (CRP)

DETAILED DESCRIPTION:
To investigate the multimodality approaches for mHSPC

ELIGIBILITY:
Inclusion Criteria:

1. Male aged ≥18 and ≤75;
2. Histologically confirmed prostate adenocarcinoma;
3. Evidence of metastasis confirmed by magnetic resonance imaging (MRI)/computed tomography (CT) scan, bone scan, or histology;
4. Clinical stage M1a (distant lymph node positive), M1b (bone metastasis), or M1c (visceral organ metastasis);
5. Prostate cancer has not received local treatment (e.g., prostate radiotherapy, cryotherapy, etc.);
6. The surgeon believes the prostate can be removed;

Exclusion Criteria:

1. The surgeon believes the disease is unresectable;
2. Life expectancy less than 2 years;
3. Active spinal cord compression;
4. History of prior local treatment for prostate cancer;
5. Difficulty swallowing, chronic diarrhea, intestinal obstruction, and other factors affecting drug intake and absorption;
6. Refusal to sign the informed consent;
7. Investigator believes the individual is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
rPFS | 3 year
  Assess how long a cancer patient lives without any signs of progression of their disease, as determined by radiographic evidence

SECONDARY OUTCOMES:
Safety of CRP in mHSPC patients | until one year after the local therapy
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Hua, M.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT06350825/Prot_ICF_000.pdf